CLINICAL TRIAL: NCT01582204
Title: Pilot Trial To Evaluate The Utility Of 124I-cG250 for The Early Detection Of Response to Therapy In Patients With Metastatic Renal Cell Carcinoma
Brief Title: Evaluate The Utility Of 124I-cG250 for The Early Detection Of Response to Therapy In Patients With Metastatic Renal Cell Carcinoma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Telix Pharmaceutical (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 11-134
Record Dates: First submitted 2012-04-18; First posted 2012-04-20 (Estimated); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Renal Cancer
Keywords: clear cell carcinoma; Kidney; MAB-124I-CG250; PET scan; CT scan; sunitinib; pazopanib; 11-134
MeSH Terms: conditions — Kidney Neoplasms; Adenocarcinoma, Clear Cell

ARMS (1):
- 124IcG250 (Experimental): This is a pilot study of 124I-cG250-PET/CT in 25 evaluable patients with advanced and/or metastatic clear cell renal cell carcinoma (ccRCC) who are scheduled to begin treatment with sunitinib or pazopanib. 124I-cG250-PET/CT will be assessed for its ability to predict response in comparison to standard CT scan of the chest, abdomen, and pelvis.
  Interventions: Drug: 124IcG250

INTERVENTIONS:
Drug: 124IcG250 — Pts will undergo baseline disease assessment with CT scans (chest, abd & pelvis), 124I-cG250-PET/CT & Tc99mMDP bone scan. W/I 7 days of their lst 124I-cG250 PET/CT, pts will start tx with sunitinib or pazopanib, dosed in successive 6-week cycles. At selected time points during the sunitinib or pazopanib cycle 1, repeat imaging with CT scan & 124I-cG250 PET/CT will be performed. After cycle 2, pts will be followed per standard of care, i.e., pts will have a standard CT scan of the chest, abd, & pelvis with contrast after cycles 2, 3, 4 & 6 (or at the time of disease progression if prior to cycle 6) for determination of best response using RECIST 1.1. Each pt will have 2 124I-cG250-PET/CT scans: baseline & week 4 (during sunitinib or pazopanib tx). All experimental imaging will take place during tx cycle 1. There will be a dosimetry sub-study for pts willing to undergo 3 additional PET/CT scans, whole body counts, & serial blood sampling, following the lst inj of 124I-cG250.

SUMMARY:
Usually, doctors monitor kidney cancer with CT scans to measure the size of tumors. Sometimes, even when a drug is working, it can take several months before the effects are seen on a regular CT scan. The purpose of this study is to see if a new kind of scan, called 124I-cG250 PET/CT, can determine response to sunitinib or pazopanib earlier than a regular CT scan.

Research has shown that certain proteins in the blood, called antibodies, can attach themselves to cancer cells without binding to normal cells. In this study, an antibody is used called chimeric G250 (cG250) that is attached to a radioactive isotope. The radioactive isotope in this study is Iodine-124 (124I). If cG250 has attached to tumors in the body, 124I shows up on the PET scan.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed clear cell carcinoma (conventional) with advanced and/or metastatic disease.
* Radiographic evidence of unidimensionally measurable disease. Lesions will be considered measurable or non- measurable as per definitions provided in RECIST version 1.1
* Subjects must be planned for treatment with approved treatment doses of a VEGF receptor TKI (e.g., sunitinib, pazopanib, cabozantinib, axitinib, sorafenib, lenvatinib).
* Male or female, 18 years of age or older.
* ECOG (Eastern Cooperative Oncology Group) performance status of ≤ 2.
* Resolution of all acute toxic effects of prior chemotherapy, radiotherapy, or surgical procedure to NCI CTCAE grade ≤2.
* The following laboratory results should be within the following limits, within 2 weeks prior to study start:
* Absolute neutrophil count (ANC) ≥1.5 x 109/L
* Total serum bilirubin <2.0 mg/dL
* Platelets ≥100,000/μL
* Serum creatinine ≤2.0 mg/dL
* Aspartate aminotransaminase (AST) ≤ 2.5 x ULN (≤ 5.0x in case of liver mets)
* Alanine aminotransferase (ALT) ≤ 2.5 x ULN (≤ 5.0x in case of liver mets)
* Valid written informed consent signed by the patient prior to any study-specific procedures.

Exclusion Criteria:

* Women who are pregnant or breast-feeding. Female patients must be surgically sterile or be postmenopausal, or must agree to use effective contraception during the period of therapy. A negative pregnancy test is required within 24 hours of administration of radiotracer and study initiation for women of childbearing age and potential.
* Other severe, acute, or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study.
* Prior treatment with a VEGF receptor TKI within a time period equivalent to 5 half-lives of the prior TKI (e.g., there should be no substantial amount of TKI remaining in the patient).
* Patient is unable to undergo contrast-enhanced CT.
* Uncontrolled or unstable hyperthyroidism or Grave's Disease.
* Contraindication to IOSATTM intake (see package insert).
* Uncontrolled active seizure disorder or history of cerebrovascular accident (CVA) or transient ischemic (TI) attack within the past 12 months.
* Unstable cardiac disease, e.g., unstable angina, congestive heart failure or myocardial infarction within the preceding 6 months.
* Known active hepatitis B/C or HIV (human immunodeficiency virus) infection.
* Prior exposure to murine proteins or chimeric antibodies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-04; Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
accuracy of predicting | 1.5 months
  The primary endpoint will be the accuracy of predicting response as per 124I-cG250- PET/CT (based on patient SUVs at day 24-29 and at day 39-42, separately) for early detection of best response to sunitinib or pazopanib as per CT imaging in patients with metastatic and/or advanced ccRCC up through 6 cycles of treatment.

SECONDARY OUTCOMES:
progression-free survival | 9 months
  Prediction of progression-free survival at 9 months as per CT imaging using SUVmax identified on 124I-cG250-PET/CT (at day 24-29).
Detection of metastatic lesions | 1 year
  Detection of metastatic lesions at baseline (number, anatomical location, size) comparing CT, PET/CT and bone scan:
  1. Number of metastases detected by CT, PET/CT and bone scan in total
  2. Number of metastases detected by CT, PET/CT and bone scan by main metastatic location (local lymph nodes, lung, bone, liver, and other)
To evaluate the radiation dosimetry of 124I-cG250. | 2 years
  using data from patients enrolled in the optional dosimetry sub-study. The data used for this purpose will include PET/CT images, whole-body counts and serum activity measurements. Results will be expressed in terms of absorbed radiation dose per unit administered activity for normal organs.

CONTACTS AND LOCATIONS:
Overall Officials: Darren Feldman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/